CLINICAL TRIAL: NCT03387969
Title: Role of CSF-CRPand Serum Procalcitonin in Differentiation Between Bacterial and Viral Meningitis in Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud abdelfattah, principal investigator, Assiut University
Other Study IDs: pediatric meningitis
Record Dates: First submitted 2017-12-24; First posted 2018-01-02 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Meningitis in Children

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — CSF analysis with culture sensitivity and gram stain .
  * CSF-CRP level measured by reagent nephelometric method by BN prospec seimense.
  * Serum procalcitonin level for all patient suspected with meningitis measured by chemilumensce on cobas E411 or by ELISA (enzyme linked immunoassay)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- meningitic group: Children suffering from fever , disturbed consciousnessand convulsion admitted in emergency department attending to assiut University Children Hospital aged between 2-18 years old
  Interventions: Procedure: CSF sample

INTERVENTIONS:
Procedure: CSF sample — for all patient CSF sample obtained for analysis , culture sensitvity and CSF-CRP.
  also blood samples will be collected and analyzed for serum procalcitonin

SUMMARY:
Meningitis is one of the major lethal infectious diseases especially for the children in developing countries .It is not always possible and often very difficult to distinguish between bacterial and viral meningitis according to CSF findings, which is not accurate 100% and leads to unnecessary antibiotic usage , So We tried to find a useful 'bedside' decision-making tool, based on laboratory results readily available at the emergency department .

DETAILED DESCRIPTION:
Meningitis, since described first in the year 1805, has been one of the major lethal infectious diseases especially for the children in developing countries .Bacterial meningitis, still one of the most life-threatening potentially serious infection worldwide of high morbidity and mortality, it is more prevalent in children and its timely and early differentiation from viral meningitis has a huge impact on the treatment of affected patients with 1.2 million cases per year, resulting in 135 000 deaths.

Case fatality rates for bacterial meningitis range from 4.5% in developed countries to 15-50% in developing countries.

A further 15-20% of survivors sustain neurological sequelae , Including presistant hearing loss and neurologic disability.

The mortality from meningitis is close to 100% in untreated individuals and can still be up to 40% in children who received appropriate antibiotic therapy in developing countries .

Most of these fatalities occur within 72 hours of admission to the hospitals. Neurological outcome and survival depends largely on damage to central nervous system prior to effective antimicrobial therapy. Quick diagnosis and effective management is the key to success . bacterial meningitis commonly caused by N.meningitis , strept.Pneumonia, H.influenza & Group B streptococci. but viral meningitis caused by Enteroviruses 50% , Herpes viruses , respiratory viruses & others itis transmitted by person to person contact through respiratory secretions or droplets.

Diagnostic dilemma is due to large spectrum of signs and symptoms and majority of children who report to hospital have already been treated with inadequate doses of antibiotics and present with atypical features of CSF examination. The only reliable method is bacterial culture of CSF which is positive only in 30-60% and it requires at least 48-72 hrs to be positive. Hence, a test that might help to diagnose and differentiate meningitis earliest is more useful to decrease expensive antibiotic for prolonged duration causing financial burden to poor parents and lengthening of hospital stay .

Hence this study will be conducted to determine and compare the sensitivity, specificity, predictive values and likelihood ratios of such laboratory tests used for diagnosing and differentiating between bacterial and viral meningitis are levels of CRP in CSF and serum procalcitonin with special reference to CSF-CRP level measured by reagent nephelometric method by BN prospec seimense, the major advantage of this method is it's rapid easy two minute reaction time . Serum procalcitonin level for all patient suspected with meningitis measured by chemilumensce on cobas E411 or by ELISA (enzyme linked immunoassay) using blood culture and gram stain as gold standard test.

.

ELIGIBILITY:
Inclusion Criteria:

* Patients at pediatric emergency care unit characterized by:

  1. Age from 2 years to 18 years old.
  2. All patients with clinical features suggestive of meningitis presented with fever, convulsions and possible meningeal signs.
  3. Immuno-compermised patients or patients on steroids specially.

Exclusion Criteria:

1. Patients above 18 years old .
2. patient with acute infections at sites other than central nervous system.
3. patients with severe hepatic dysfunction .
4. patient with positive family history of metabolic disease .
5. patients known to had congenital CNS abnormality.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children at pediatric emergency care unit attending to Assuit University Children Hospital Aged from 2 years to 18 years old presented with fever, convulsions, disturbed consciousness and possible meningeal sign
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2019-01-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
differentiation between bacterial and viral meningitis | 12 month
  by using simple bed side diagnostic test as CSF-CRP and procalcitonin confirmed by CSF culture sensitivity and CSF analysis with gram stain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tankhiwale SS, Jagtap PM, Khadse RK, Jalgaonkar SV. Bacteriological study of pyogenic meningitis with special reference to C-reactive protein. Indian J Med Microbiol. 2001 Jul-Sep;19(3):159-60. PMID 17664824
- [Background] Antona D, Leveque N, Chomel JJ, Dubrou S, Levy-Bruhl D, Lina B. Surveillance of enteroviruses in France, 2000-2004. Eur J Clin Microbiol Infect Dis. 2007 Jun;26(6):403-12. doi: 10.1007/s10096-007-0306-4. PMID 17534678
- [Background] Konstantinidis T, Cassimos D, Gioka T, Tsigalou C, Parasidis T, Alexandropoulou I, Nikolaidis C, Kampouromiti G, Constantinidis T, Chatzimichael A, Panopoulou M. Can Procalcitonin in Cerebrospinal Fluid be a Diagnostic Tool for Meningitis? J Clin Lab Anal. 2015 May;29(3):169-74. doi: 10.1002/jcla.21746. Epub 2014 May 5. PMID 24797775
- [Background] Anh DD, Riewpaiboon A, Tho le H, Kim SA, Nyambat B, Kilgore P. Treatment costs of pneumonia, meningitis, sepsis, and other diseases among hospitalized children in Viet Nam. J Health Popul Nutr. 2010 Oct;28(5):436-42. doi: 10.3329/jhpn.v28i5.6151. PMID 20941894
- [Background] -Amol R. Shinde1, K. S. Ghorpade2, A. M. Siddiqui1. A study of Cerebrospinal Fluid Adenosine deaminase and C-reactive protein in Bacterial, Tubercular and Viral meningitis. Asian Journal of Biomedical and Pharmaceutical Sciences, 2015; 5(44): 15-18
- [Background] -Patel N, Patel U, Nagpal AC, Jain RK. Evaluating Utility of C reactive protein in Differentiating Bacterial from Non-Bacterial Meningitis in Tertiary Care Hospital, in Central India . International Journal of Medical Research and Review. April-June, 2013/ Vol 1/ Issue 2
- [Background] Quagliarello VJ, Scheld WM. Treatment of bacterial meningitis. N Engl J Med. 1997 Mar 6;336(10):708-16. doi: 10.1056/NEJM199703063361007. No abstract available. PMID 9041103
- [Background] Muller B, White JC, Nylen ES, Snider RH, Becker KL, Habener JF. Ubiquitous expression of the calcitonin-i gene in multiple tissues in response to sepsis. J Clin Endocrinol Metab. 2001 Jan;86(1):396-404. doi: 10.1210/jcem.86.1.7089. PMID 11232031
- [Background] Bergallo M, Costa C, Margio S, Sidoti F, Terlizzi ME, Cavallo R. Development of a multiplex polymerase chain reaction for detection and typing of major human herpesviruses in cerebrospinal fluid. Can J Microbiol. 2007 Oct;53(10):1117-22. doi: 10.1139/w07-074. PMID 18026203
- [Background] Big C, Reineck LA, Aronoff DM. Viral infections of the central nervous system: a case-based review. Clin Med Res. 2009 Dec;7(4):142-6. doi: 10.3121/cmr.2009.864. Epub 2009 Nov 4. PMID 19889944
- [Background] DeBiasi RL, Kleinschmidt-DeMasters BK, Weinberg A, Tyler KL. Use of PCR for the diagnosis of herpesvirus infections of the central nervous system. J Clin Virol. 2002 Jul;25 Suppl 1:S5-11. doi: 10.1016/s1386-6532(02)00028-8. PMID 12091076
- [Background] Chen DY, Chen YM, Ho WL, Chen HH, Shen GH, Lan JL. Diagnostic value of procalcitonin for differentiation between bacterial infection and non-infectious inflammation in febrile patients with active adult-onset Still's disease. Ann Rheum Dis. 2009 Jun;68(6):1074-5. doi: 10.1136/ard.2008.098335. No abstract available. PMID 19435724
- [Background] Hofer N, Zacharias E, Muller W, Resch B. An update on the use of C-reactive protein in early-onset neonatal sepsis: current insights and new tasks. Neonatology. 2012;102(1):25-36. doi: 10.1159/000336629. Epub 2012 Apr 11. PMID 22507868
- [Background] Christ-Crain M, Muller B. Procalcitonin in bacterial infections--hype, hope, more or less? Swiss Med Wkly. 2005 Aug 6;135(31-32):451-60. doi: 10.4414/smw.2005.11169. PMID 16208582
- [Background] Mary R, Veinberg F, Couderc R. [Acute meningitidis, acute phase proteins and procalcitonin]. Ann Biol Clin (Paris). 2003 Mar-Apr;61(2):127-37. French. PMID 12702467
- [Background] Tunkel AR, Hartman BJ, Kaplan SL, Kaufman BA, Roos KL, Scheld WM, Whitley RJ. Practice guidelines for the management of bacterial meningitis. Clin Infect Dis. 2004 Nov 1;39(9):1267-84. doi: 10.1086/425368. Epub 2004 Oct 6. No abstract available. PMID 15494903
- [Background] Leveque N, Van Haecke A, Renois F, Boutolleau D, Talmud D, Andreoletti L. Rapid virological diagnosis of central nervous system infections by use of a multiplex reverse transcription-PCR DNA microarray. J Clin Microbiol. 2011 Nov;49(11):3874-9. doi: 10.1128/JCM.01214-11. Epub 2011 Sep 14. PMID 21918017